CLINICAL TRIAL: NCT07303686
Title: Pilot Study to Assess De-escalation of Ustekinumab Therapy in Patients With Crohn's Disease and Ulcerative Colitis
Brief Title: De-escalation of Ustekinumab Therapy in Patients With Crohn's Disease and Ulcerative Colitis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Janssen Inc. (Industry)
Responsible Party: Principal Investigator, waqqas.afif, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-5567
Record Dates: First submitted 2025-10-02; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Crohn Disease (CD); Ulcerative Colitis (UC)
Keywords: CD; UC; ustekinumab; UST
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative | interventions — Ustekinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ustekinumab Q4w (Other)
  Interventions: Biological: Ustekinumab 90 mg SC q8w
- Ustekinumab Q8w (Other)
  Interventions: Biological: Ustekinumab 90 mg SC q12w

INTERVENTIONS:
Biological: Ustekinumab 90 mg SC q8w — Sub-group switching from Q4w to Q8w
  Arms: Ustekinumab Q4w
Biological: Ustekinumab 90 mg SC q12w — Sub-group switching from Q8w to Q12w
  Arms: Ustekinumab Q8w

SUMMARY:
The goal of this clinical trial is to evaluate whether disease remission can be maintained when biologic therapy is reduced in patients with Crohn"s disease (CD) and ulcerative colitis (UC) taking ustekinumab (UST).

The main question it aims to answer is:

Can we de-escalate UST subcutaneous dose either from every 4 weeks (Q4) to every 8 weeks (Q8) or every 8 weeks (Q8) to every 12 weeks (Q12) in CD or UC patients in deep remission without loosing their response? Researchers will follow UST blood levels, inflammation markers and intestinal mucosa integrity and to see if UST dose can be reduced while maintaining clinical remission.

Participants will:

Change UST dosing from Q4 to Q8 or from Q8 to Q12. Visit the clinic once every 12 weeks for checkups and tests.

DETAILED DESCRIPTION:
Participation in this research study will last 12 months and will include 4-6 visits.

ELIGIBILITY:
Inclusion Criteria:

* Clinical remission
* Biochemical remission
* Endoscopy remission
* Not on corticosteroid
* A woman must be ;
* not of childbearing potential
* of childbearing potential and practicing a medically accepted method of contraception.
* Able t provide informed consent

Exclusion Criteria:

* On more than one biologics drug
* Use of oral or topical steroids within 6months of study entry
* pregnancy
* Any issue that could lead to non-compliance, as alcohol, drug use
* Unable to provide consent or t comply with follw-up visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Loss of clinical remission | From treatment switch to end of participation (12 months)
  Proportion of patients experiencing loss of remission

SECONDARY OUTCOMES:
Time-to-loss of Remission | From treatment switch to end of participation (12 months)
Change from Baseline in the C-reactive protein (CRP) level at loss of remission. | 12 months
  To define if CRP level is a predictor of loss of remission.
Change from Baseline in the calprotectin level at loss of remission. | 12 months
  To define if calprotectin level is a predictor of loss of remission.
Disease duration before loss of remission. | Up to 50 years.
  Define if disease duration is a predictor of loss of remission.
Change in drug concentration before loss of remission. | 12 months
  Define if drug concentration in blood is a predictor of loss of remission.

CONTACTS AND LOCATIONS:
Locations (1):
- MUHC - Montreal General Hospital, Montreal, Quebec, Canada